CLINICAL TRIAL: NCT03297294
Title: A Double-blind, Placebo-controlled, Randomized Trial to Determine the Safety and Efficacy of EMA401 in Reducing 24-hour Average Pain Intensity Score in Patients With Painful Diabetic Neuropathy (EMPADINE)
Brief Title: Safety and Efficacy of EMA401 in Patients With Painful Diabetic Neuropathy (PDN)
Acronym: EMPADINE
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Study was terminated due to animal toxicity data
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CEMA401A2202; 2016-000281-39 (EudraCT Number)
Record Dates: First submitted 2017-09-26; First posted 2017-09-29 (Actual); Results first posted 2020-06-04 (Actual); Last update posted 2021-10-08 (Actual); Status verified 2021-10

CONDITIONS: Painful Diabetic Neuropathy
Keywords: Painful diabetic neuropathy; Neuropathic pain; Angiotensin II type 2 receptor antagonist; adult; EMA401; diabetic neuropathy
MeSH Terms: conditions — Diabetic Neuropathies; Neuralgia | interventions — EMA400

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- EMA401 (Experimental): During the treatment epoch, patients will receive EMA401 for 12 weeks. During the treatment withdrawal epoch, patients will receive EMA401 or matching placebo for 1 week.
  Interventions: Drug: EMA401; Drug: Placebo
- Placebo (Placebo Comparator): Participants will receive matching placebo to EMA401 during both the treatment and treatment withdrawal epochs for a total of 13 weeks.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: EMA401 — capsules, oral
  Arms: EMA401
Drug: Placebo — Placebo to EMA401 capsules, oral

SUMMARY:
The purpose of this study is to evaluate safety and efficacy of EMA401 compared to placebo in patients with painful diabetic neuropathy (PDN).

DETAILED DESCRIPTION:
This was an interventional, randomized, parallel, placebo-controlled, double-blind treatment study consisting of 3 periods i.e. Screening, Treatment, and Treatment withdrawal. Patients were planned to be randomized in a 1:1 ratio to Placebo b.i.d. or EMA401 100 mg b.i.d.. Concomitant use of pregabalin or duloxetine at stable doses was allowed. Based on historical data, it was planned that the study would enroll approximately 50% of patients who were on stable doses of concomitant pregabalin or duloxetine in the study. At the end of treatment period the 100mg b.i.d. arm was re-randomized (1:1) to the same treatment or placebo. Placebo arm stayed on placebo. The planned duration of treatment period was 12 weeks and 1 week of treatment withdrawal at the end of treatment period.

The study was terminated early due to pre-clinical toxicity data that became available after start of trial. Novartis implemented a Urgent Safety Measure (USM) which instructed sites to discontinue study treatment immediately and to have all patients return for additional laboratory assessments (full hematology including coagulation and clinical chemistry panel). Safety data from the USM was presented as a separate outcome measure table and not included in the Adverse Event section

ELIGIBILITY:
Inclusion Criteria:

* At the time of Screening, must have had documented diagnosis of Type I OR Type II diabetes mellitus (DM) with painful distal symmetrical sensorimotor neuropathy (ICD-10 code G63.2) of more than 6 months duration with any one or more of the following:

  * Neuropathic symptoms (e.g. numbness, non-painful paresthesias or tingling, non-painful sensory distortions or misinterpretations, etc.)
  * Decreased distal sensation (e.g. decreased vibration, pinprick sensation, light touch, etc.)
* Been assessed as suffering from moderate to severe neuropathic pain across the Screening epoch (NRS ≥ 4).
* A score of ≥4 on the Douleur Neuropathique en 4 Questions (DN4) questionnaire at Screening.

Exclusion Criteria:

* Women of child-bearing potential, defined as all women physiologically capable of becoming pregnant, unless they were using highly effective methods of contraception during dosing and for 3 days after stopping of study medication. Highly effective contraception methods included:

  * Total abstinence (when this was is in line with the preferred and usual lifestyle of the subject). Periodic abstinence (e.g., calendar, ovulation, symptothermal, post-ovulation methods) and withdrawal were not acceptable methods of contraception.
  * Female sterilization (have had surgical bilateral oophorectomy with or without hysterectomy), total hysterectomy or tubal ligation at least six weeks before taking investigational drug. In case of oophorectomy alone, only when the reproductive status of the woman had been confirmed by follow up hormone level assessment.
  * Male sterilization (at least 6 months prior to screening). For female subjects on the study, the vasectomized male partner should have been the sole partner for that subject.
  * Placement of an intrauterine device (IUD) or intrauterine system (IUS).
* History or current diagnosis of electrocardiogram (ECG) abnormalities indicating significant risk of safety for patients participating in the study.
* Major depressive episode within 6 months prior to Screening and/or a history of diagnosed recurrent major depressive disorder according to Diagnostic and Statistical Manual of Mental Disorders, 5th Edition (DSM-V) diagnostic criteria.
* Had evidence of significant renal insufficiency or pre-existing liver condition.
* Had platelets ≤ 100 x 10^9/L, or neutrophil count < 1.2 x 10^9/L (or equivalent), hemoglobin ≤ 100 g/L for women or hemoglobin ≤ 110 g/L for men.
* Participants whose glycemic control had been unstable within 3 months immediately prior to screening (e.g., ketoacidosis requiring hospitalization, any recent episode of hypoglycemia requiring assistance through medical intervention, uncontrolled hyperglycemia)
* Patients who had any differential diagnosis of PDN including but not limited to other neuropathies (e.g. Vitamin B12 deficiency, Chronic Inflammatory Demyelinating Polyneuropathy), polyradiculopathies, central disorders (e.g. demyelinating disease), or rheumatological disease (e.g., foot arthritis, plantar fasciitis).
* Patient was unwilling or unable to complete daily eDiary.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 142 (Actual)
Dates: Start 2018-03-14 (Actual); Primary Completion 2019-03-25 (Actual); Study Completion 2019-03-25 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (59):
- Australia (4):
  - Novartis Investigative Site, Broadmeadow, New South Wales
  - Novartis Investigative Site, Orange, New South Wales
  - Novartis Investigative Site, Adelaide, South Australia
  - Novartis Investigative Site, Heidelberg Heights, Victoria
- Austria (3):
  - Novartis Investigative Site, Graz
  - Novartis Investigative Site, Klagenfurt
  - Novartis Investigative Site, Vienna
- Belgium (3):
  - Novartis Investigative Site, Edegem
  - Novartis Investigative Site, Liège
  - Novartis Investigative Site, Pellenberg
- Bulgaria (2):
  - Novartis Investigative Site, Sofia, Sofia-Grad
  - Novartis Investigative Site, Sofia
- Canada (4):
  - Novartis Investigative Site, Ontario, CAN
  - Novartis Investigative Site, Thornhill, Ontario
  - Novartis Investigative Site, Toronto, Ontario
  - Novartis Investigative Site, Laval, Quebec
- Denmark (3):
  - Novartis Investigative Site, Aarhus
  - Novartis Investigative Site, Gentofte Municipality
  - Novartis Investigative Site, Odense C
- Novartis Investigative Site, Tampere, Finland
- Novartis Investigative Site, Boulogne-Billancourt, France
- Germany (8):
  - Novartis Investigative Site, Bielefeld
  - Novartis Investigative Site, Düsseldorf
  - Novartis Investigative Site, Essen
  - Novartis Investigative Site, Halle
  - Novartis Investigative Site, Kassel
  - Novartis Investigative Site, Kiel
  - Novartis Investigative Site, Leipzig
  - Novartis Investigative Site, Wiesbaden
- Hungary (8):
  - Novartis Investigative Site, Debrecen, HUN
  - Novartis Investigative Site, Esztergom, HUN
  - Novartis Investigative Site, Szeged, HUN
  - Novartis Investigative Site, Balatonfüred
  - Novartis Investigative Site, Budapest
  - Novartis Investigative Site, Kistarcsa
  - Novartis Investigative Site, Pécs
  - Novartis Investigative Site, Szeged
- Novartis Investigative Site, Oslo, Norway
- Poland (3):
  - Novartis Investigative Site, Krakow, POL
  - Novartis Investigative Site, Bialystok
  - Novartis Investigative Site, Warsaw
- Portugal (6):
  - Novartis Investigative Site, Caldas da Rainha
  - Novartis Investigative Site, Lisbon
  - Novartis Investigative Site, Matosinhos Municipality
  - Novartis Investigative Site, Porto
  - Novartis Investigative Site, Viana do Castelo
  - Novartis Investigative Site, Vila Nova de Gaia
- Slovakia (3):
  - Novartis Investigative Site, Lučenec, Slovak Republic
  - Novartis Investigative Site, Bratislava
  - Novartis Investigative Site, Prešov
- Spain (2):
  - Novartis Investigative Site, Seville, Andalusia
  - Novartis Investigative Site, Madrid
- United Kingdom (7):
  - Novartis Investigative Site, Bradford, West Yorkshire
  - Novartis Investigative Site, Bath
  - Novartis Investigative Site, Bournemouth
  - Novartis Investigative Site, Edinburgh
  - Novartis Investigative Site, London
  - Novartis Investigative Site, Middlesbrough
  - Novartis Investigative Site, Oldham

IPD SHARING:
Plan to Share IPD: Undecided
Novartis is committed to sharing with qualified external researchers, access to patient-level data and supporting clinical documents from eligible studies. These requests are reviewed and approved by an independent review panel on the basis of scientific merit. All data provided is anonymized to respect the privacy of patients who have participated in the trial in line with applicable laws and regulations.
  This trial data availability is according to the criteria and process described on www.clinicalstudydatarequest.com.

REFERENCES:
- [Derived] Rice ASC, Dworkin RH, Finnerup NB, Attal N, Anand P, Freeman R, Piaia A, Callegari F, Doerr C, Mondal S, Narayanan N, Ecochard L, Flossbach Y, Pandhi S. Efficacy and safety of EMA401 in peripheral neuropathic pain: results of 2 randomised, double-blind, phase 2 studies in patients with postherpetic neuralgia and painful diabetic neuropathy. Pain. 2021 Oct 1;162(10):2578-2589. doi: 10.1097/j.pain.0000000000002252. PMID 33675631
- See also: A Plain Language Trial Summary is available on novartisclinicaltrials.com — https://www.novctrd.com/ctrdweb/patientsummary/patientsummaries?patientSummaryId=619

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Three hundred six patients were screened and 137 randomized
Groups:
- EMA401 100mg BID DB: Ema401 100 mg was administered orally twice a day during double blind (DB) treatment period
- Placebo BID DB: Matching placebo capsules administered orally twice a day during double blind (DB) treatment period
- EMA401 100mg BID -> EMA401 100mg BID TW; EMA401 100mg BID -> Placebo BID TW: Participants on EMA401 100mg were randomized 1:1 to EMA401 100mg or placebo at end of DB treatment period (week 12)
- Placebo BID -> Placebo BID TW: Participants on placebo remained on placebo at end of DB treatment period (week 12)
Period: Double-Blind Treatment Period (DB)
Arm/Group | EMA401 100mg BID DB | Placebo BID DB | EMA401 100mg BID -> EMA401 100mg BID TW | EMA401 100mg BID -> Placebo BID TW | Placebo BID -> Placebo BID TW
Started | 70 | 67 | 0 | 0 | 0
Completed (Study completers completed the treatment phase regardless of completion of study treatment.) | 32 | 30 | 0 | 0 | 0
Not Completed | 38 | 37 | 0 | 0 | 0
Not completed — Study terminated by sponsor | 30 | 31 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 4 | 4 | 0 | 0 | 0
Not completed — Adverse Event | 3 | 1 | 0 | 0 | 0
Not completed — Physician Decision | 1 | 1 | 0 | 0 | 0
Period: Treatment Withdrawal Period (TW)
Arm/Group | EMA401 100mg BID DB | Placebo BID DB | EMA401 100mg BID -> EMA401 100mg BID TW | EMA401 100mg BID -> Placebo BID TW | Placebo BID -> Placebo BID TW
Started | 0 | 0 | 14 | 12 | 27
Completed | 0 | 0 | 14 | 11 | 27
Not Completed | 0 | 0 | 0 | 1 | 0
Not completed — Study terminated by sponsor | 0 | 0 | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | EMA401 100mg BID DB | Placebo BID DB | Total
Number analyzed (Participants) | 70 | 67 | 137
Age, Customized [Count of Participants; unit: Participants]
  18 - 64 years | 34 | 33 | 67
  65 - 84 years | 36 | 33 | 69
  ≥ 85 years | 0 | 1 | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 20 | 24 | 44
  Male | 50 | 43 | 93
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Caucasian | 70 | 63 | 133
  Asian | 0 | 1 | 1
  Other | 0 | 3 | 3
Body mass index [Median (Full Range); unit: kg/m^2] | 30.8 [22.7 to 43.2] | 30.2 [19.5 to 48.2] | 30.6 [19.5 to 48.2]

OUTCOME MEASURES:

1. Primary Outcome: Change in Weekly Mean 24-hour Average Pain Score Using the 11 Point Numerical Rating Scale (NRS) From Baseline to Week 12
Description: The NRS is an 11-point scale ranging from zero ("no pain") to ten ("pain as bad as you can imagine") for self-reporting of pain by patients. The following parameters were evaluated using the 11-point NRS: 24-hour Average Pain Score and 24-hour Worst Pain Score Patients evaluated their "average pain" and "worst pain" during the past 24 hours in the evening prior to sleep by touching the appropriate corresponding number between zero and ten on a eDiary device.
Time Frame: Baseline up to Week 12
Population: Full analysis set
Measure: Least Squares Mean (Standard Error); unit: scores on a scale
Arm/Group | EMA401 100mg BID DB | Placebo BID DB
Number analyzed (Participants) | 70 | 67
scores on a scale
  Week 4 | -1.0 (0.21) | -0.8 (0.18)
  Week 8 | -1.7 (0.29) | -1.1 (0.26)
  Week 12 | -1.9 (0.31) | -1.3 (0.27)
Statistical Analysis 1: Comparison: EMA401 100mg BID DB vs Placebo BID DB; Test type: Superiority — at week 12; p = 0.101, ANCOVA; least squares mean = -0.6, 95% CI 2-sided [-1.4 to 0.1], Standard Error of Mean 0.39

2. Secondary Outcome: Change in Neuropathic Pain Symptom Inventory (NPSI) From Baseline to Week 12
Description: The Neuropathic Pain Symptom Inventory (NPSI) is a 12 item patient reported outcome measure that contains 10 descriptors representing 5 dimensions of pain (burning pain, deep/pressing pain, paroxysmal pain, evoked pain and paraesthesia/dysesthesia) and 2 temporal items designed to assess pain duration and the number of pain paroxysms. The sum of the responses to the 10 questions (all except temporal questions) was regarded as the total score and was divided by 10 (10 questions). The range of the total score and of the 5 dimensional scores is 0 to 10. Lower values represent better outcomes.
Time Frame: Baseline up to Week 12
Measure: Least Squares Mean (Standard Error); unit: scores on a scale
Arm/Group | EMA401 100mg BID DB | Placebo BID DB
Number analyzed (Participants) | 70 | 67
scores on a scale
  Week 4 | -1.2 (0.19) | -1.0 (0.18)
  Week 8 | -1.3 (0.25) | -0.9 (0.22)
  Week 12 | -1.6 (0.32) | -1.1 (0.26)
Statistical Analysis 1: Comparison: EMA401 100mg BID DB vs Placebo BID DB; At week 12; Test type: Superiority; p = 0.168, ANCOVA; LS mean difference = -0.5, 95% CI 2-sided [-1.3 to 0.2], Standard Error of Mean 0.38

3. Secondary Outcome: Change in Brief Pain Inventory-Short Form Interference (BPI-SF) Mean Total Score From Baseline to Week 12
Description: The BPI-SF is a validated, self-administered (at clinic) questionnaire that assesses pain severity and its mpact on daily functions. Patients were asked to complete the 7-item pain interference scale that assessed the degree to which pain interfered with walking and other physical activity, work, mood, relations with others and sleep using a zero to ten scale with zero being "does not interfere" and ten being "completely interferes". The BPI total score is the sum of the 7 items. Each item ranges from 0 to 10, thus the total score ranges from 0 to 70. Lower values indicate a better outcome.
Time Frame: Baseline up to Week 12
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | EMA401 100mg BID DB | Placebo BID DB
Number analyzed (Participants) | 70 | 67
scores on a scale | -12.03 (13.336) | -10.83 (14.602)

4. Secondary Outcome: Change in Weekly Mean of the 24-hour Worst Pain Score, Using an 11-point NRS, From Baseline to Week 12
Description: as for outcome 1
Time Frame: Baseline up to Week 12
Measure: Mean (Standard Deviation); unit: scores on numeric rating scale
Arm/Group | EMA401 100mg BID DB | Placebo BID DB
Number analyzed (Participants) | 70 | 67
scores on numeric rating scale | -1.63 (1.837) | -1.28 (1.577)

5. Secondary Outcome: Number of Participants Per Patient Global Impression of Change Category at Week 12
Description: The Patient Global Impression of Change (PGIC) is a patient-reported instrument that measures change in overall status on a scale ranging from one ("very much improved") to seven ("very much worse"). The PGIC is based on the validated Clinical Global Impression of Change scale. The PGIC was to be completed by patients using the electronic tablet at the site
Time Frame: Baseline up to Week 12
Measure: Count of Participants; unit: Participants
Arm/Group | EMA401 100mg BID DB | Placebo BID DB
Number analyzed (Participants) | 70 | 67
Participants
  Very much improved | 4 | 2
  Much improved | 7 | 11
  Minimally improved | 17 | 18
  No change | 18 | 14
  Minimally worse | 3 | 2
  Much worse | 0 | 0
  Very much worse | 0 | 0
  Missing | 21 | 20

6. Secondary Outcome: Percentage of Patients Achieving at Least 30% Pain Reduction at Week 12 on NRS 11 Point Scale
Description: The NRS is an 11-point scale ranging from zero ("no pain") to ten ("pain as bad as you can imagine") for self-reporting of pain by patients. The number of patients with observed response, i.e. a decrease of 30% units in weekly mean of the 24-hour average pain score NRS. Logistic regression model with region, treatment, sex, use of PHN medications (yes/no) as factors and age and baseline NRS as covariates. An odds ratio >1 = higher chance of a clinically important improvement.
Time Frame: Baseline up to Week 12
Population: Full analysis set
Measure: Number; unit: % of participants - model adjusted rate
Arm/Group | EMA401 100mg BID DB | Placebo BID DB
Number analyzed (Participants) | 70 | 67
% of participants - model adjusted rate
  Week 4 - at least 30% pain reduction: number analyzed (Participants) | 18 | 14
  Week 4 - at least 30% pain reduction | 34.0 | 24.7
  Week 12 - at least 30% pain reduction: number analyzed (Participants) | 14 | 12
  Week 12 - at least 30% pain reduction | 52.7 | 40.4
Statistical Analysis 1: Comparison: EMA401 100mg BID DB vs Placebo BID DB; Week 12; Test type: Superiority; p = 0.255, Regression, Logistic; Odds Ratio (OR) = 1.6, 95% CI 2-sided [0.7 to 3.9]

7. Secondary Outcome: Percentage of Patients Achieving at Least 50% Pain Reduction at Week 12 on NRS 11 Point Scale
Description: The NRS is an 11-point scale ranging from zero ("no pain") to ten ("pain as bad as you can imagine") for self-reporting of pain by patients. The number of patients with observed response, i.e. a decrease of 50% units in weekly mean of the 24-hour average pain score NRS. Logistic regression model with region, treatment, sex, use of PHN medications (yes/no) as factors and age and baseline NRS as covariates. An odds ratio >1 = higher chance of a clinically important improvement.
Time Frame: Baseline up to Week 12
Population: Full analysis set
Measure: Number; unit: % of participants - model adjusted rate
Arm/Group | EMA401 100mg BID DB | Placebo BID DB
Number analyzed (Participants) | 70 | 67
% of participants - model adjusted rate | 31.4 | 14.1
Statistical Analysis 1: Comparison: EMA401 100mg BID DB vs Placebo BID DB; Test type: Superiority; p = 0.100, Regression, Logistic; Odds Ratio (OR) = 2.8, 95% CI 2-sided [0.8 to 9.6]

8. Secondary Outcome: Mean Change in Insomnia Severity Index (ISI) From Baseline to Week 12
Description: Patients were asked to complete the ISI using five-point Likert-style scale as a measure of perceived sleep difficulties. The questionnaire assessed the severity of insomnia, satisfaction with current sleep pattern, sleep interference, "noticeability" of sleeping problem to others and concern about sleeping problems. The scale consists of 7 items. The sum of seven items represents the total score. Each of the 7 items is scored using a range from 0 to 4, thus the total score values ranges from zero to 28. Lower values represent better outcomes.
Time Frame: Baseline up to Week 12
Population: Full analysis set
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | EMA401 100mg BID DB | Placebo BID DB
Number analyzed (Participants) | 70 | 67
scores on a scale | -4.00 (4.854) | -1.03 (6.312)

9. Secondary Outcome: Plasma Pharmacokinetics (PK) Concentrations at Week 8 and 12
Description: Due to the premature termination of the study, the number of patients and observations providing PK data was much smaller than planned, and no PK model was developed. As a consequence, no PK parameters (Cmax, Tmax, AUC) were derived for this study. Only, summary statistics of the plasma concentrations were calculated
Time Frame: Week 8 (Prior dose, 1-3 hours, 4-6 hours), Week 12 (Prior dose, 1-3 hours, 4-6 hours)
Population: PK analysis set
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | EMA401 100mg BID DB
Number analyzed (Participants) | 32
ng/mL
  Week 8 Prior dose | 30.5 (126.6)
  Week 8 1-3 hours | 205.1 (212.8)
  Week 8 4-6 hours | 72.8 (115.2)
  Week 12 Prior dose: number analyzed (Participants) | 25
  Week 12 Prior dose | 29.5 (209.3)
  Week 12 1-3 hours: number analyzed (Participants) | 26
  Week 12 1-3 hours | 118.4 (278.3)
  Week 12 4-6 hours: number analyzed (Participants) | 26
  Week 12 4-6 hours | 89.8 (117.0)

10. Secondary Outcome: Percentage of Patients Who Required Rescue Medication in Double-blind Treatment Period
Description: Patients were allowed to take acetaminophen/paracetamol up to a maximum of 3 g daily (divided into 4 times/day) for unacceptable pain due to any reason during the study. This medication use was to be recorded in eDiary prior to use. Percentages of patients presented are those who required rescue meds within 7 days prior to visit.
Time Frame: Baseline and weekly up to 12 weeks, once during double-blind period
Population: Full analysis set
Measure: Number; unit: Percentage of participants
Arm/Group | EMA401 100mg BID DB | Placebo BID DB
Number analyzed (Participants) | 70 | 67
Percentage of participants
  Week 1 | 13.0 | 10.6
  Week 2 | 7.7 | 9.5
  Week 4 | 8.6 | 7.0
  Week 6 | 7.8 | 7.5
  Week 8 | 9.3 | 9.5
  Week 10 | 5.3 | 13.2
  Week 12 | 2.9 | 8.6
  At least once during double-blind period | 20.0 | 19.4

11. Secondary Outcome: Percentage of Patients Who Required Rescue Medication in Treatment Withdrawal Period
Description: as for outcome 10
Time Frame: Week 12 to Week 13 (planned duration subject to varibility in visit scheduling)
Population: Full analysis set
Measure: Number; unit: Percentage of participants
Arm/Group | EMA401 100mg BID -> EMA401 100mg BID TW | EMA401 100mg BID -> Placebo BID TW | Placebo BID -> Placebo BID TW
Number analyzed (Participants) | 35 | 35 | 67
Percentage of participants | 14.3 | 8.3 | 7.4

12. Secondary Outcome: Time to First Rescue Medication Intake
Description: Patients were allowed to take acetaminophen/paracetamol up to a maximum of 3 g daily (divided into 4 times/day) for unacceptable pain due to any reason during the study. This medication use was to be recorded in eDiary prior to use. Patients who did not take any rescue medication were censored at the last date of double-blind treatment period.
Time Frame: Baseline up to day 92
Population: Full analysis set
Measure: Median (Full Range); unit: days
Arm/Group | EMA401 100mg BID DB | Placebo BID DB
Number analyzed (Participants) | 70 | 67
days | 44.0 [2 to 90] | 56.5 [2 to 92]

13. Secondary Outcome: Treatment Emergent Adverse Events During Urgent Safety Measure (USM) Follow-Up
Description: Participants were instructed to stop taking drug immediately upon termination of study and asked to come in for two unscheduled visits for follow up safety assessments
Time Frame: Approximately from 3 weeks after end of study up to 16 weeks
Population: The Overall Number of Participants Analyzed reflects the Safety population, regardless of whether they completed the study
Measure: Count of Participants; unit: Participants
Arm/Group | EMA401 100mg BID -> EMA401 100mg BID TW | EMA401 100mg BID -> Placebo BID TW | Placebo BID -> Placebo BID TW
Number analyzed (Participants) | 34 | 35 | 66
Participants
  Peritoneal adhesions | 1 | 0 | 0
  Cholelithiasis | 1 | 0 | 0
  Liver abscess | 1 | 0 | 0
  Blood creatinine increased | 0 | 0 | 1

ADVERSE EVENTS:
Time Frame: Adverse events were collected from first dose of study treatment until end of study treatment plus 21 days post treatment, up to maximum duration of 111 days
Description: Any sign or symptom that occurs during the study treatment plus the 21 days post treatment are reported in adverse event (AE) section. Upon termination of study, participants were instructed to attend two unscheduled visits for follow-up safety assessments for Urgent Safety Measure (USM) follow-up. Adverse events collected during USM are not included in this AE section but reported in secondary outcome measure 13 entitled Treatment Emergent Adverse Events During Urgent Safety Measure Follow-up
Arm/Group | EMA401 100mg BID DB | Placebo BID DB | EMA401 100mg BID -> EMA401 100mg BID TW | EMA401 100mg BID -> Placebo BID TW | Placebo BID -> Placebo BID TW
All-Cause Mortality (participants affected / at risk) | 0/69 | 0/66 | 0/14 | 0/12 | 0/26
Serious Adverse Events (participants affected / at risk) | 5/69 | 3/66 | 0/14 | 0/12 | 0/26
Other Adverse Events (participants affected / at risk) | 23/69 | 10/66 | 1/14 | 2/12 | 0/26
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | EMA401 100mg BID DB (N=69) | Placebo BID DB (N=66) | EMA401 100mg BID -> EMA401 100mg BID TW (N=14) | EMA401 100mg BID -> Placebo BID TW (N=12) | Placebo BID -> Placebo BID TW (N=26)
Acute coronary syndrome (Cardiac disorders) | 0 | 1 | 0 | 0 | 0
Product intolerance (General disorders) | 1 | 0 | 0 | 0 | 0
Cholecystitis acute (Hepatobiliary disorders) | 2 | 0 | 0 | 0 | 0
Cholelithiasis (Hepatobiliary disorders) | 1 | 0 | 0 | 0 | 0
Erysipelas (Infections and infestations) | 0 | 1 | 0 | 0 | 0
Localised infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | EMA401 100mg BID DB (N=69) | Placebo BID DB (N=66) | EMA401 100mg BID -> EMA401 100mg BID TW (N=14) | EMA401 100mg BID -> Placebo BID TW (N=12) | Placebo BID -> Placebo BID TW (N=26)
Palpitations (Cardiac disorders) | 0 | 1 | 0 | 1 | 0
Abdominal pain upper (Gastrointestinal disorders) | 5 | 0 | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 4 | 1 | 0 | 0 | 0
Nasopharyngitis (Infections and infestations) | 4 | 6 | 0 | 0 | 0
Gamma-glutamyltransferase increased (Investigations) | 4 | 1 | 0 | 0 | 0
Lipase increased (Investigations) | 6 | 0 | 1 | 0 | 0
Headache (Nervous system disorders) | 4 | 4 | 0 | 0 | 0
Hypertension (Vascular disorders) | 1 | 2 | 0 | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (ie, data from all sites) in the clinical trial.

DOCUMENTS (2):
  • Study Protocol (2017-09-15): https://cdn.clinicaltrials.gov/large-docs/94/NCT03297294/Prot_001.pdf
  • Statistical Analysis Plan (2019-06-18): https://cdn.clinicaltrials.gov/large-docs/94/NCT03297294/SAP_000.pdf